CLINICAL TRIAL: NCT01086748
Title: A Phase 2, Multicenter, Double-Blind, Placebo-Controlled Comparator Study of 2 Doses of LY2140023 Versus Placebo in Patients With DSM-IV-TR Schizophrenia
Brief Title: A Study in Schizophrenia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11958; H8Y-MC-HBBM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; LY 2140023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 160 mg LY2140023 (Experimental): 80 mg LY2140023 administered orally, twice daily (BID) for up to 7 weeks.
  Interventions: Drug: LY2140023
- 4 mg Risperidone (Active Comparator): 2 mg risperidone administered orally, BID for up to 7 weeks.
  Interventions: Drug: Risperidone
- Placebo (Placebo Comparator): Placebo administered orally, BID for up to 7 weeks.
  Interventions: Drug: Placebo
- 80 mg LY2140023 (Experimental): 40 mg LY2140023 administered orally, BID for up to 7 weeks.
  Interventions: Drug: LY2140023

INTERVENTIONS:
Drug: Risperidone — Administered orally.
  Arms: 4 mg Risperidone
Drug: Placebo — Administered orally.
  Arms: Placebo
Drug: LY2140023 — Administered orally.
  Arms: 160 mg LY2140023; 80 mg LY2140023

SUMMARY:
An inpatient/outpatient study to see if LY2140023 is better than placebo in acutely ill patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR; APA 2000) (Disorganized, 295.10; Catatonic, 295.20; Paranoid 295.30; or Undifferentiated, 295.90) and confirmed by the Structured Clinical Interview for DSM-IV-TR (SCID).
* Non pregnant female patients who agree to use acceptable birth control
* At entry to the study must be considered moderately ill in the opinion of the investigator
* Willing to participate in a minimum of 3 weeks of inpatient hospitalization and this must be appropriate for the patient in the clinical judgment of the investigator.
* 1 year history of Schizophrenia prior to entering the study
* At study entry patients with a history of antipsychotic treatment must have a lifetime history of at least one hospitalization for the treatment of schizophrenia, not including the hospitalization required for study. Patients who have never taken antipsychotic treatment may enter the study even without a history of hospitalization.
* At study entry patients with a history of antipsychotic treatment must have a history of at least one episode of illness exacerbation requiring an intensification of treatment intervention or care in the last 2 years, not including the present episode of illness. Patients who have never taken antipsychotic treatment may enter the study without a past history of illness exacerbation and intensification of treatment in the last 2 years.
* At study entry patients must have experienced an exacerbation of illness within the 2 weeks prior to entering the study, leading to an intensification of psychiatric care in the opinion of the investigator. If exacerbation occurs in patients who are presently hospitalized, the patient must not have been hospitalized longer than 60 days at entry of the study

Exclusion Criteria:

* Participated in any clinical trial with any pharmacological treatment intervention for which they received a study-related medication in the 6 months prior to visit 1
* Previously completed or withdrawn from this study, or any other study investigating LY2140023 or any predecessor molecules with glutamatergic activity.
* Treatment with clozapine at doses greater than 200 mg daily within 12 months prior to entering the study, or who have received any clozapine at all during the month before entering the study
* Patients currently receiving treatment (within 1 dosing interval, minimum of 4 weeks, prior entering the study) with a depot formulation of an antipsychotic medication.
* Patients who are currently suicidal.
* Females who are pregnant, nursing, or who intend to become pregnant within 30 days of completing the study.
* Patients with uncorrected narrow-angle glaucoma, uncontrolled diabetes, certain diseases of the liver, renal insufficiency, uncontrolled thyroid condition or other serious or unstable illnesses
* Have a history of one or more seizures, except for those who experienced a single simple febrile seizure between ages 6 months and 5 years
* Patients are excluded if their, biological father, mother, brother, sister, or child has a history of idiopathic epilepsy.
* Within 1 year of study enrollment, patients have a history of central nervous system infection, uncontrolled migraine, transient ischemic attack (TIA), or head trauma with loss of consciousness or a post-concussive
* Patients are excluded if they have a lifetime history of any of the following:

  * head trauma, stroke, or CNS infection with persistent neurological deficit (focal or diffuse);
  * brain surgery;
  * an electroencephalogram with paroxysmal (epileptiform) activity, or
  * brain structural lesion, including developmental abnormalities, as determined by examination or previous neuroimaging studies that are consistent with a diagnosable neurological disease or syndrome.
* Electroconvulsive therapy (ECT) within 3 months of entering the study or who will have ECT at any time during the study.
* Leukopenia
* Medical history of Human Immunodeficiency Virus positive (HIV+) status.
* Higher than normal blood prolactin levels
* Certain electrocardiogram results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
A change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score in overall schizophrenia population | baseline, up to 7 weeks of treatment
A change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score in a genetic subgroup of schizophrenia patients | baseline, up to 7 weeks of treatment

SECONDARY OUTCOMES:
A change from baseline in the Personal and Social Performance (PSP) score in the overall schizophrenia population | baseline, up to 7 weeks of treatment
A change from baseline in the Personal and Social Performance (PSP) score in a genetic subgroup of schizophrenia patients | baseline, up to 7 weeks of treatment
A change from baseline in the PANSS positive scale | baseline, up to 7 weeks of treatment
A change from baseline in the PANSS negative scale | baseline, up to 7 weeks of treatment
A change from baseline in PANSS General Psychopathology subscale | baseline, up to 7 weeks of treatment
A change from baseline in the Clinical Global Impression-Severity Scale (CGI-S) | baseline, up to 7 weeks of treatment
A change from baseline in the 16-item Negative Symptoms Assessment (NSA-16) | baseline, up to 7 weeks of treatment
A change from baseline in the Montgomery-Ǻsberg Depression Rating Scale (MADRS) | baseline, up to 7 weeks of treatment
PANSS total score | up to 7 weeks of treatment
A change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score in a female patients | baseline, up to 7 weeks of treatment
Rate of discontinuation | baseline, up to 7 weeks of treatment
Time to discontinuation | baseline, up to 7 weeks of treatment
A change from baseline on the EuroQol - 5 Dimensions (EQ-5D) Questionnaire | baseline, up to 7 weeks of treatment
A change from baseline on resource utilization, as measured by the Schizophrenia Resource Use Model (S-RUM) | Baseline up to 7 weeks of treatment
A change from baseline on functional capacity, as measured by the Subjective Well-Being Under Neuroleptic Treatment Scale - Short Form (SWN-S) | baseline, up to 7 weeks of treatment
A change from baseline in Barnes Akathisia Scale (BAS) | baseline, up to 7 weeks of treatment
A change from baseline in Simpson-Angus Scale (SAS) | baseline, up to 7 weeks of treatment
A change from baseline in Abnormal Involuntary Movement Scale (AIMS) | baseline, up to 7 weeks of treatment
A mean change from baseline in Prolactin levels | baseline, up to 7 weeks of treatment
A change from baseline in weight | baseline, up to 7 weeks of treatment
Number of Treatment Emergent Adverse Events (TEAEs) | Up to 7 weeks of treatment
Change from baseline in electrocardiogram parameters | baseline, up to 7 weeks of treatment
A change from baseline in neurological examination | baseline, up to 7 weeks of treatment
Statistically different changes in vital signs from baseline | baseline, up to 7 weeks of treatment
Statistically different changes in lab values from baseline | baseline, up to 7 weeks of treatment
Population pharmacokinetics (PK) of LY2140023 | baseline, up to 7 weeks of treatment
A change from baseline in Columbia- Suicide Severity Rating Scale (C-SSRS) | baseline, up to 7 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paramount, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Creve Coeur, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeSoto, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb, Croatia
- Russia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Khot'kovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lipetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nizhny Novgorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Samara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl

REFERENCES:
- [Derived] Kinon BJ, Millen BA, Zhang L, McKinzie DL. Exploratory analysis for a targeted patient population responsive to the metabotropic glutamate 2/3 receptor agonist pomaglumetad methionil in schizophrenia. Biol Psychiatry. 2015 Dec 1;78(11):754-62. doi: 10.1016/j.biopsych.2015.03.016. Epub 2015 Mar 19. PMID 25890643
- [Derived] Downing AM, Kinon BJ, Millen BA, Zhang L, Liu L, Morozova MA, Brenner R, Rayle TJ, Nisenbaum L, Zhao F, Gomez JC. A Double-Blind, Placebo-Controlled Comparator Study of LY2140023 monohydrate in patients with schizophrenia. BMC Psychiatry. 2014 Dec 10;14:351. doi: 10.1186/s12888-014-0351-3. PMID 25539791